CLINICAL TRIAL: NCT03453086
Title: A Randomized Controlled Study Comparing Thoracic Paravertebral Block to Serratus Anterior Plane Block in Breast Surgery
Brief Title: Comparison of Thoracic Paravertebral Block , Pectoral Nerve Block to Serratus Anterior Plane Block in Breast Surgery, A Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Mohamed, Ahmed A., M.D. (Individual); Laila Halim Doss (Unknown); Ahmed Zaghloul Fouad (Unknown); Michael Zarif Sobhy (Unknown)
Responsible Party: Principal Investigator, Ahmed Abdalla, Assistant Professor of Anesthesia &I.C.U and Pain Clinic, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N19-2016/MD
Record Dates: First submitted 2017-12-29; First posted 2018-03-05 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Comparison of Thoracic Paravertebral Block to Serratus Anterior Plane Block in Breast Surgery
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: Although thoracic epidural analgesia is the gold standard technique after breast surgery paravertebral block (PVB) has become a potential alternative approach. However, both techniques may be associated with serious complications such as pneumothorax, total spinal anaesthesia and inadvertent intravascular injection. Recently since the advent of ultrasound (US) in anaesthetic practice several interfascial plane blocks have been described. Serratus plane block is a novel interfascial plane block which can provide analgesia after breast surgery.
  The serratus anterior plane block is an interfascial plane block where the local anaesthetics are injected superficial to serratus anterior at the 5th rib level in the mid axillary line. The serratus plane block is a progression from Blanco's et al work with the Pecs I and II blocks by making the technique easier in its application using single injection and to lower the potential side-effects
Who Masked: Participant, Care Provider
Masking Description: •Patients will be randomly allocated to one of the two groups by sealed closed envelop technique
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I: (Active Comparator): These patients will receive single ipsilateral Ultrasound TPVB which performed with the patient in the sitting position at the level of the T4 with the probe in a vertical position 2.5-3 cm lateral to the midline. The midpoint of the transducer is to be placed in a longitudinal paramedian plane between two transverse processes which visualized with the superior costo-transverse ligament and the pleura visible in between . After this, 15-20 cc of bupivacaine 0.25% will be injected
  Interventions: Procedure: Thoracic paravertebral block(TPVB) group
- Group II : (Active Comparator): These patients will receive serratus anterior plane block. The block will be performed while the patient is in the supine position by using a linear Ultrasound probe of high frequency (6-13 MHz) after sheathing. The probe will be placed over the mid-clavicular region of the thoracic cage in a sagittal plane. The ribs will be counted inferiorly and laterally, until the 5th rib is identified in the midaxillary line. The latissimus dorsi (superficial and posterior) , teres major (superior) and serratus muscles (deep and inferior) will be then easily identifiable by U/S overlying the fifth rib.
  Interventions: Procedure: Thoracic paravertebral block(TPVB) group

INTERVENTIONS:
Procedure: Thoracic paravertebral block(TPVB) group — Thoracic paravertebral block group (TPVB) group: The midpoint of the transducer is to be placed in a longitudinal paramedian plane between two transverse processes.Tuohy needle will be introduced in a cephalad direction. The tip of the needle will be advanced under direct visualization until it pierces the superior costo-transverse ligament. When the needle tip is located immediately above the pleura, the needle is aspirated to confirm the absence of blood or air.
  Serratus anterior plane block group (SAP) group: The US probe will be placed over the mid-clavicular region of the thoracic cage in a sagittal plane. The ribs will be counted until the 5th rib is identified in the midaxillary line. The latissimus dorsi, teres major and serratus muscles will be then easily identifiable by US overlying the fifth rib. The needle will be introduced in-plane with respect to the US probe from supero-anterior to postero-inferior
  Other Names: Serratus anterior plane block( SAP) group

SUMMARY:
The investigators hypothesize that the analgesic efficacy of ultrasound-guided serratus anterior plane block will provide better analgesia with fewer complications in comparison to ultrasound guided thoracic paravertebral block

DETAILED DESCRIPTION:
•The blocks techniques:

* Group I: Thoracic paravertebral block group (TPVB group n=15) These patients will receive single ipsilateral ultrasound-guided thoracic paravertebral block. TPVB will be performed with the patient in the sitting position at the level of the 4th thoracic vertebra under complete aseptic precaution with the probe in a vertical position approximately 2.5-3 cm lateral to the midline. The midpoint of the transducer is to be placed in a longitudinal paramedian plane between two transverse processes. Both transverse processes should be visualized, with the superior costo-transverse ligament and the pleura visible in between .An 18-20 gauge Tuohy needle will be introduced in a cephalad direction. The tip of the needle will be advanced under direct visualization until it pierces the superior costo-transverse ligament. the investigators will inject small aliquots of normal saline intermittently as the investigators advance the needle to confirm the position of the tip. When the needle tip is located immediately above the pleura, the needle is aspirated to confirm the absence of blood or air. After this, 15-20 cc of bupivacaine 0.25% will be injected. Spread of local anaesthetic with depression of the pleura will be clearly visualized. The extent of local anaesthetic spread should be evaluated by moving the ultrasound probe superiorly and inferiorly.
* Group II :Serratus anterior plane block group (SAP group n= 15) These patients will receive serratus anterior plane block. The SAP block will be performed while the patient is in the supine position by using a linear US probe of high frequency (6-13 MHz) after sheathing. The probe will be placed over the mid-clavicular region of the thoracic cage in a sagittal plane. The ribs will be counted inferiorly and laterally, until the 5th rib is identified in the midaxillary line. The latissimus dorsi (superficial and posterior), teres major (superior) and serratus muscles (deep and inferior) will be then easily identifiable by ultrasound overlying the fifth rib. The needle (Stimuplex, B Braun, Germany 22-G, 50-mm) will be introduced in-plane with respect to the ultrasound probe from supero-anterior to postero-inferior. Under continuous ultrasound guidance, the investigators will inject 20 cc of bupivacaine 0.25%. The sensory level will be tested with pin prick and ice pack before induction of general anesthesia

ELIGIBILITY:
Inclusion Criteria:

1. Female patients
2. Breast surgery with or without axillary clearance.
3. Age from 20 to 60 years.
4. ASA I, II, III.

Exclusion Criteria:

1. Major reconstructive breast surgery.
2. Age younger than 20 or older than 60 years.
3. ASA IV, V.
4. Hypersensitivity to any drug to be used.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-12 (Actual)

PRIMARY OUTCOMES:
First pain medication request | 24 hours
  Time to the first pain medication request till application of the block

SECONDARY OUTCOMES:
Time of pain onset | 24 hours
  Time of onset of Pain
Hemodynamics (heart rate) | 24 hours
  Hemodynamics in the form of heart rate "beats per minute"
Hemodynamics (ABP) | 24 hours
  Hemodynamics in the form of arterial blood pressure" mm Hg".
Nausea and vomiting | 24 hours
  Postoperative nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdalla, M.D, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Ahmed Abdalla Mohamed, Cairo
  - Kasr Alainy Hospitals, Cairo

IPD SHARING:
Plan to Share IPD: No
Via scholar Gate